CLINICAL TRIAL: NCT00862446
Title: Use of Omega-3 Fat Emulsion (Omegaven) in Infants With Parenteral Nutrition Associated Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080887
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Parenteral Nutrition Associated Liver Disease
Keywords: Parenteral nutrition associate liver disease; TPN cholestasis; TPN Associated Liver Disease
MeSH Terms: interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): All infants will receive Omegaven
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — 1 gram/kg/day daily until on feeds

SUMMARY:
Babies in the newborn intensive care unit who are dependent upon intravenous nutrition for a long period of time frequently develop liver damage. The fat used is called intralipid and is made from soybean oil. There is a suggestion in the literature that using fish oil based fats called omega-3 fat emulsions can decrease or even reverse this liver damage. We will offer babies with evidence of liver damage and no ability to eat,the Omegaven and see if the liver damage reverses.

DETAILED DESCRIPTION:
Babies in the newborn intensive care unit with evidence of liver damage from Total Parenteral Nutrition (TPN), as indicated by a direct bilirubin of greater than 2.5 , and who will not be fed for at least another month will be offered the trial. they will be changed from the intralipid to Omegaven as the source of their fat. We will continue routine monitoring of their nutrition and liver function.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the newborn intensive care unit
* TPN cholestasis of at least 2.5 mg/dl
* Anticipated TPN treatment for at least one month
* signed informed consent

Exclusion Criteria:

* Enrollment in another trial
* Lack of consent

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Monroe Carell Jr Children's Hospital at vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Omegaven Treatment: All participants received Omegaven: 1 gram/kg/day daily until they were able to ingest adequate nutrition enterally
Period: Overall Study
Arm/Group | Omegaven Treatment
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omegaven Treatment
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: days] | 63.875 (32.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 48
Direct Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 6.25 (3.83)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resolution of the Direct Hyperbilirubinemia
Description: Defined as direct bilirubin <2.0 mg/dL
Time Frame: At discharge or up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven Treatment
Number analyzed (Participants) | 48
Participants | 29

ADVERSE EVENTS:
Time Frame: Baseline to Week 10
Description: The only adverse collected were mortality, coagulopathy, hypertriglyceridemia
Arm/Group | Omegaven Treatment
All-Cause Mortality (participants affected / at risk) | 6/48
Serious Adverse Events (participants affected / at risk) | 5/48
Other Adverse Events (participants affected / at risk) | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omegaven Treatment (N=48)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) — Prolonged or excessive bleeding
Hypertriglyceridemia (Blood and lymphatic system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT00862446/Prot_SAP_000.pdf